CLINICAL TRIAL: NCT00652301
Title: A Randomized, Double-Blind, Placebo-Controlled,4-Period, Crossover Study to Evaluate the Effects of Ezetimibe and Simvastatin, Coadministered and Alone, on Intestinal Absorption of Cholesterol
Brief Title: A Research Study to Evaluate MK0653 (Ezetimibe) and Simvastatin, Given Together and Alone, on Intestinal Absorption of Cholesterol (0653-050)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 0653-050; MK0653-050; 2007_559
Record Dates: First submitted 2008-03-31; First posted 2008-04-03 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Cholesterol
MeSH Terms: interventions — Ezetimibe; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Experimental): ezetimibe 10 mg tablet plus simvastatin 20 mg tablet
  Interventions: Drug: ezetimibe; Drug: simvastatin
- 2 (Active Comparator): ezetimibe 10 mg tablet
  Interventions: Drug: ezetimibe; Drug: Comparator: Placebo (unspecified)
- 3 (Active Comparator): simvastatin 20 mg tablet
  Interventions: Drug: Comparator: Placebo (unspecified); Drug: simvastatin
- 4 (Placebo Comparator): matching placebo
  Interventions: Drug: Comparator: Placebo (unspecified)

INTERVENTIONS:
Drug: ezetimibe — ezetimibe 10 mg tablet. Duration of Treatment 31 Weeks.
  Other Names: MK0653
  Arms: 1; 2
Drug: Comparator: Placebo (unspecified) — matching placebo tablet. Duration of Treatment 31 Weeks.
  Arms: 2; 3; 4
Drug: simvastatin — simvastatin 20 mg tablet. Duration of Treatment 31 Weeks.
  Other Names: MK0733
  Arms: 1; 3

SUMMARY:
To determine the effect of ezetimibe and simvastatin given together, and ezetimibe and simvastatin given alone on intestinal cholesterol absorption.

DETAILED DESCRIPTION:
Patients will be randomized into 1 of 4 treatment sequences involving 4 consecutive 7-week treatment periods.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males between the ages of 18-55 with LDL More than 130, but less than 180

Exclusion Criteria:

* Individuals with drug or substance abuse
* Individuals with poor mental function
* Individuals having more than 14 alcoholic drinks a week
* Individuals that have been treated with any other investigational drug in the last 30 days

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2003-07; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
reduced intestinal cholesterol absorption with ezetimibe + simvastatin vs simvastatin alone. | Based on 7 week treatment periods.

SECONDARY OUTCOMES:
To determine the effects of ezetimibe alone and simvastatin alone on intestinal cholesterol absorption. | Based on 7 week treatment periods.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Sudhop T, Reber M, Tribble D, Sapre A, Taggart W, Gibbons P, Musliner T, von Bergmann K, Lutjohann D. Changes in cholesterol absorption and cholesterol synthesis caused by ezetimibe and/or simvastatin in men. J Lipid Res. 2009 Oct;50(10):2117-23. doi: 10.1194/jlr.P900004-JLR200. Epub 2009 Apr 20. PMID 19380898